CLINICAL TRIAL: NCT04662294
Title: Clinical Trial for the Safety and Efficacy of CD 70 CAR T for Patients With CD70 Positive Malignant Hematologic Diseases
Brief Title: CD 70 CAR T for Patients With CD70 Positive Malignant Hematologic Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD70-001
Record Dates: First submitted 2020-10-22; First posted 2020-12-10 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2020-12

CONDITIONS: Acute Myeloid Leukemia; Non-hodgkin's Lymphoma; Multiple Myeloma
Keywords: CAR T-cell therapy; CD70; Acute Myeloid Leukemia; Non-Hodgkin's lymphoma; Multiple Myeloma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T-ALL (Experimental)
  Interventions: Biological: CD70 CAR T-cells
- T-NHL (Experimental)
  Interventions: Biological: CD70 CAR T-cells
- AML (Experimental)
  Interventions: Biological: CD70 CAR T-cells

INTERVENTIONS:
Biological: CD70 CAR T-cells — Each subject receive CD70 CAR T-cells by intravenous infusion
  Other Names: CD70 CAR-T cells injection

SUMMARY:
A Study of CD 70 CAR T for patients with CD70 positive malignant hematologic diseases

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study. This study is indicated for CD 70 CAR T for patients with CD70 positive malignant hematologic diseases. The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products. 108 patients will be enrolled. Primary objective is to explore the safety,main consideration is dose-related safety.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria only for AML:

1. Histologically confirmed diagnosis of CD70 AML per the US National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Acute Myeloid Leukemia (2016.v1);
2. Relapsed or refractory CD70+ AML (meeting one of the following conditions):

   1. CR not achieved after standardized chemotherapy;
   2. CR achieved following the first induction, but CR duration is less than 12 months;
   3. Ineffectively after first or multiple remedial treatments;
   4. 2 or more relapses;
3. The number of primordial cells in bone marrow is > 5% (by morphology), and/or > 0.01% (by flowcytometry);
4. Total bilirubin ≤ 51 umol/L, ALT and AST ≤ 3 times of upper limit ofnormal, creatinine ≤ 176.8 umol/L;
5. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥50%;
6. No active infection in the lungs, blood oxygen saturation in indoorair is ≥ 92%;
7. Estimated survival time ≥ 3 months;
8. ECOG performance status 0 to 2;
9. Patients or their legal guardians volunteer to participate in the studyand sign the informed consent.

Inclusion criteria only for NHL:

1. No gender and age limit;
2. Histologically confirmed diagnosis of DLBCL (NOS), FL, DLBCL transformed from CLL/SLL, PMBCL, and HGBCL per the WHO Classification Criteria for Lymphoma (2016);
3. Relapsed or refractory CD70+ NHL (meeting one of the following conditions):

   1. No response or relapse after second-line or above chemotherapy regimens;
   2. Primary drug resistance;
   3. Relapse after auto-HSCT;
4. At least one assessable tumor lesion per Lugano 2014 criteria

Inclusion criteria only for MM:

1. Histologically confirmed diagnosis of CD70 multiple myeloma (MM)：

   1. According to the diagnostic criteria of IMWG multiple myeloma, the diagnosis was recurrent / refractory multiple myeloma
   2. Cases with recurrent positive minimal residual disease;
   3. Extramedullary leision which is hard to be eradicated by chemotherapy or radiotherapy.
2. No gender and age limit;
3. Total bilirubin ≤ 51 umol/L, ALT and AST ≤ 3 times of upper limit of normal, creatinine ≤ 176.8 umol/L;
4. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥50%;
5. No active infection in the lungs, blood oxygen saturation in indoorair is ≥ 92%;
6. Estimated survival time ≥ 3 months;
7. ECOG performance status 0 to 2;
8. Patients or their legal guardians volunteer to participate in the studyand sign the informed consent.

Common inclusion criteria :

1. Total bilirubin ≤ 51 umol/L, ALT and AST ≤ 3 times of upper limit of normal, creatinine ≤ 176.8 umol/L;
2. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥ 50%;
3. No active infection in the lungs, blood oxygen saturation in indoor air is ≥ 92%;
4. Estimated survival time ≥ 3 months;
5. ECOG performance status 0 to 2;
6. Patients or their legal guardians volunteer to participate in the study and sign the informed consent -

Exclusion Criteria:

1. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases;
2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
3. Pregnant (or lactating) women;
4. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
5. Active infection of hepatitis B virus or hepatitis C virus;
6. Concurrent therapy with systemic steroids within 2 weeks prior to screening, except for the patients recently or currently receiving inhaled steroids;
7. Previously treated with any CAR-T cell product or other geneticallymodified T cell therapies;
8. Creatinine >2.5mg/dl, or ALT / AST>3 times of normal amounts, or bilirubin>2.0 mg/dl;
9. Other uncontrolled diseases that were not suitable for this trial;
10. Patients with HIV infection;
11. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study. -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-11-18 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CD70 targeted CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after CD70 targeted CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Acute Myeloid Leukemia (AML), Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi) at Month 1, 3, 6, 12, 18 and 24
AML, Overall survival (OS) | Up to 2 years after CD70 CAR-T cells infusion
  From the first infusion of CD70 CAR-T cells to death or the last visit
AML, Event-free survival (EFS) | Up to 2 years after CD70 CAR-T cells infusion
  From the first infusion of CD70 CAR-T cells to the occurrence of any event, including death, relapse or gene relapse, disease progression (any one occurs first), and the last visit
Non-Hodgkin's lymphoma (NHL), Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi) at Month 1, 3, 6, 12, 18 and 24
NHL, Overall survival (OS) | Up to 2 years after CD70 CAR-T cells infusion
  From the first infusion of CD70 CAR-T cells to death or the last visit
NHL, Event-free survival (EFS) | Up to 2 years after CD70 CAR-T cells infusion
  From the first infusion of CD70 CAR-T cells to the occurrence of any event, including death, relapse or gene relapse,
Multiple myeloma (MM), Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi) at Month 1, 3, 6, 12, 18 and 24
MM, Overall survival (OS) | Up to 2 years after CD70 CAR-T cells infusion
  From the first infusion of CD70 CAR-T cells to death or the last visit
MM, Event-free survival (EFS) | Up to 2 years after CD70 CAR-T cells infusion
  From the first infusion of CD70 CAR-T cells to the occurrence of any event, including death, relapse or gene relapse
Quality of life | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale [For item1-28: max score: 112, min score: 28, higher scores mean a better outcome; for item 28-29: max score: 14, min score: 2, higher scores mean a worse outcome] to measure Quality of life at Baseline, Month 1, 3, 6, 9 and 12
Activities of Daily Living (ADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Activities of Daily Living (ADL) scale (Barthel Index) [max score: 100, min score: 0, higher scores mean a better outcome] at Baseline, Month 1, 3, 6, 9 and 12
Instrumental Activities of Daily Living (IADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Instrumental Activities of Daily Living (IADL) scale [max score: 56, min score: 14, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12
Hospital Anxiety and Depression Scale (HADS) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Hospital Anxiety and Depression Scale (HADS) [max score: 42, min score: 0, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dewulf J, Flieswasser T, Delahaye T, Vangestel C, Miranda A, de Haard H, Jacobs J, Smits E, Van den Wyngaert T, Elvas F. Site-specific 68Ga-labeled nanobody for PET imaging of CD70 expression in preclinical tumor models. EJNMMI Radiopharm Chem. 2023 Apr 24;8(1):8. doi: 10.1186/s41181-023-00194-3. PMID 37093350
- [Derived] Golubovskaya V. CAR-T Cells Targeting Immune Checkpoint Pathway Players. Front Biosci (Landmark Ed). 2022 Apr 2;27(4):121. doi: 10.31083/j.fbl2704121. PMID 35468680